CLINICAL TRIAL: NCT00539721
Title: A Randomized, Double-Blind, Double-Dummy, Dose-Ranging, Active- and Placebo-Controlled Study of Single-Dose Oral Rolapitant Monotherapy for the Prevention of Postoperative Nausea and Vomiting (PONV)
Brief Title: A Randomized Controlled Study of Rolapitant for the Prevention of Nausea and Vomiting Following Surgery (Study P04937AM1)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P04937
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Nausea; Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Rolapitant Dose 1 (Experimental)
  Interventions: Drug: Rolapitant Dose 1
- Rolapitant Dose 2 (Experimental)
  Interventions: Drug: Rolapitant Dose 2
- Rolapitant Dose 3 (Experimental)
  Interventions: Drug: Rolapitant Dose 3
- Rolapitant Dose 4 (Experimental)
  Interventions: Drug: Rolapitant Dose 4
- Ondansetron (Active Comparator)
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rolapitant Dose 1 — Rolapitant 5 mg (4 capsules) x 1 oral and ondansetron placebo x 1 intravenous on Day 1
  Arms: Rolapitant Dose 1
Drug: Rolapitant Dose 2 — Rolapitant 20 mg (4 capsules) x 1 oral and ondansetron placebo x 1 intravenous on Day 1
  Arms: Rolapitant Dose 2
Drug: Rolapitant Dose 3 — Rolapitant 70 mg (4 capsules) x 1 oral and ondansetron placebo x 1 intravenous on Day 1
  Arms: Rolapitant Dose 3
Drug: Rolapitant Dose 4 — 200 mg (4 capsules) x 1 oral and ondansetron placebo x 1 intravenous on Day 1
  Arms: Rolapitant Dose 4
Drug: Ondansetron — Ondansetron 4 mg x 1 intravenous and rolapitant placebo (4 capsules) x 1 oral on Day 1
  Arms: Ondansetron
Drug: Placebo — Rolapitant placebo (4 capsules) x 1 oral and ondansetron placebo x 1 intravenous on Day 1
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, controlled study in women who are having elective open abdominal surgery with general anesthesia and who are expected to need patient-controlled analgesia (PCA) after surgery. The primary objective is to assess the effect of rolapitant in the prevention of postoperative nausea and vomiting as measured by the prevention of vomiting in the first 24 hours after surgery. Participation in the study may last up to 3 months. The total duration of the study will be approximately 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older of any race with an American Society of Anesthesiologists (ASA) physical status of I to III who are scheduled to undergo elective open abdominal surgery under general anesthesia.
* Women whose postoperative hospitalization is expected to last at least 24 hours
* Women expected to require postoperative intravenous opioid PCA.
* Women whose surgery is expected to require at least 1 hour, but not more than 4 hours, of general anesthesia using the regimen defined in this protocol.
* Women of childbearing potential who have a negative pregnancy test or women who have been surgically sterilized or are postmenopausal.

Exclusion Criteria:

* Women with clinically significant or unstable cardiac, respiratory, hepatic, renal, or other major organ system disease.
* Women with a known hypersensitivity to ondansetron (or any other 5-HT3 antagonist), to any agent that is part of the anesthesia regimen, or to other medications to be administered under this protocol.
* Women who are scheduled to undergo certain types of surgery.
* Women who are breastfeeding.
* Women who have retching/vomiting or moderate or severe nausea in the 24 hours prior to surgery or suffer from chronic nausea and/or vomiting.
* Women with a body mass index (BMI) >40.
* Women who have participated in a clinical trial of an investigational drug within 30 days prior to drug administration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
No emetic episodes regardless of rescue medication use. | First 24 hours after surgery.